CLINICAL TRIAL: NCT02738372
Title: The Influence of Biopsychosocial Factors and Peripheral and/or Central Sensitization in Predicting the Recovery of Chronic Shoulder Pain: a Prospective Cohort Study. Study Protocol
Brief Title: Influence of Biopsychosocial Factors and Central Sensitization in Predicting the Recovery of Chronic Shoulder Pain
Status: Completed | Type: Observational
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Other Study IDs: UMalaga
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2018-10

CONDITIONS: Chronic Shoulder Pain
Keywords: Chronic Pain; Biopsychosocial Factors; Shoulder pain; Prognosis; Central Nervous System Sensitization
MeSH Terms: conditions — Chronic Pain; Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Shoulder Pain: 1. Men / women aged between 18 and 70 years.
  2. Patients suffering from shoulder pain, defined as pain presented or exacerbated by movements in the shoulder, pain intensity ≥ 2 measured by a numerical scale with values from 0 to 10, meaning 0= no pain and 10= the worst pain, will be included in this study, among all these following shoulder pain conditions: (i) Rotator Cuff tendinopathy; (ii) Adhesive Capsulitis; (iii) glenohumeral instability; (iv) SLAP lesion; (v) and/or acromioclavicular pathology. Subjects will not be required to undergo diagnostic imaging (i.e. Magnetic Resonance Imaging) to diagnosis the pathology because of the recruitment will be carried out by clinical findings.
  3. Duration of symptoms: greater than 3 months.
  Interventions: Other: Diagnosis/Prognosis

INTERVENTIONS:
Other: Diagnosis/Prognosis — The present study will be a 24 months multi-center, triple-blind, prospective, cohort study which will be carried out between April 2016 and March 2018. Subjects diagnosed of rotator cuff (RC) tendinopathy, adhesive capsulitis (AC), glenohumeral instability, SLAP lesion, and/or acromioclavicular pathology and fulfill the inclusion criteria will be asked for participating in our study. Several questionnaires that will test the influence of different biopsychosocial factors and the presence of Central Sensitization will be administrated to these subjects. The outcomes will be assessed at baseline and 5 follow-ups (after 3, 6, 12, 18 and 24 months, t1-t6).

SUMMARY:
Background: Shoulder pain is the third most common musculoskeletal condition presenting to physicians or physiotherapists ) in primary healthcare after low back and neck pain being a significant cause of morbidity and functional disability in both working and general population. Despite the large group of individuals seeking for primary care services, about 50% of patients with shoulder pain still report persistent pain after 12-18 months. As a result, socio-economic burdens are considerable due to extensive use of heath care services, sickness absence, disability pension, and loss of productivity as well as, patient´s suffering.

Aims: the primary aim of this study was to evaluate what biopsychosocial factors predict a better and/or poor outcome in patients with Chronic shoulder pain. The secondary aim was to analyze the role of central sensitization in predicting a better and/or poor outcome in patients with Chronic shoulder pain.

Hypothesis:

1. A high level of physical inactivity, kinesiophobia, fear avoidance and pain catastrophizing and low level of self-efficacy will ease the perpetuation of Chronic shoulder pain.
2. The presence of central sensitization will predict a poor outcome in patients with chronic shoulder pain.

DETAILED DESCRIPTION:
The present study will be a 24 months multi-center, double-blind, prospective, cohort study which will be carried out between April 2016 and March 2018. Subjects diagnosed of rotator cuff (RC) tendinopathy, adhesive capsulitis (AC), glenohumeral instability, superior labrum anterior to posterior (SLAP) lesion, and/or acromioclavicular pathology and fulfill the inclusion criteria will be asked for participating in the investigators study. Several questionnaires that will test the influence of different biopsychosocial factors and the presence of Central Sensitization will be administrated to these subjects. The outcomes will be assessed at baseline and 5 follow-ups (after 3, 6, 12, 18 and 24 months, t1-t6).

Subjects will attend for their routine clinical appointment. The examiners will carry out the clinical consultation according to usual practice. Subjects who fulfill the selection criteria will be asked whether they wish to be considered for trial participation. Examiners will inform subjects who are interested in participation. Ineligible subjects and those who do not wish to participate in the trial will receive normal clinical care delivered by clinicians according to the best clinical practice.

Anonymized age, gender and visual analogue scale (VAS)- verbal numeric rating scale (VNRS) for pain will be collected for those subjects who decline to take part in the project, in order to assess the external validity of the recruited sample of subjects.

Eligible patients who are interested in the trial will be asked to provide written informed consent to participate. The examiners will allocate the participants in an unique study group. Participants will then complete several questionnaires at baseline, 3, 6, 12, 18 and 24 months after the beginning of the study. A blinded examiner will deliver these questionnaires. Subsequent sessions will occur at the follow-up visits. Participants will be asked about any problems they had had during the previous months before following-up. There will be brief discussion about whether participants have subjected for any treatment (physical, pharmacological, injection and/or no treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Men / women aged between 18 and 70 years.
2. Patients suffering from shoulder pain, defined as pain presented or exacerbated by movements in the shoulder, pain intensity = 2 measured by a numerical scale with values from 0 to 10, meaning 0= no pain and 10= the worst pain, will be included in this study, among all these following shoulder pain conditions: (i) rotator cuff (RC) tendinopathy ; (ii) adhesive capsulitis (AC) ; (iii) glenohumeral instability ; (iv) SLAP lesion; (v) and/or acromioclavicular pathology. Subjects will not be required to undergo diagnostic imaging (i.e MRI) to diagnosis the pathology because of the recruitment will be carried out by clinical findings.
3. Duration of symptoms: greater than 3 months.

Exclusion Criteria:

1. Recent shoulder dislocation (1 year prior) and/or systemic diseases such as rheumatoid arthritis, osteoarthritis, fibromyalgia and/or polymyalgia rheumatica.
2. Shoulder pain considered to be originated in the cervical region and other traumas or if there is a neurological dysfunction (i.e multiple sclerosis), osteoporosis, hemophilia and / or cancer.
3. Inability to provide informed consent and/or complete written questionnaires.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects between 18-70 years with chronic shoulder pain
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-11; Primary Completion 2019-11 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline The brief pain inventory short form (BIP-SF) at 3,6,12,18 and 24 months | Pain will be evaluated at baseline and 5 follow-ups (3,6,12,18 and 24 months).
  Pain will be assessed with The brief pain inventory short form (BIP-SF). This will be used to assess how pain interferes with patient's functioning in addition to measuring the intensity and location of pain.

SECONDARY OUTCOMES:
Change from baseline Pain catastrophizing at 3, 6, 12, 18 and 24 months assessed with The Pain Catastrophizing Scale (PSC) | Pain catastrophizing will be evaluated at baseline and 5 follow-ups (3,6,12,18 and 24 months).
  The catastrophic thinking bout pain will be assessed with The Pain Catastrophizing Scale (PSC).
Change from baseline Kinesiophobia at 3,6,12,18 and 24 months assessed with Tampa Scale For Kinesiophobia (TSK) | Kinesiophobia will be evaluated at baseline and 5 follow-ups (3,6,12,18 and 24 months).
  The fear of movement (kinesiophobia) will be assessed with Tampa Scale For Kinesiophobia (TSK).
Change from baseline Fear avoidance at 3,6,12,18 and 24 months assessed with Fear Avoidance Belief Questionnaire (FABQ) | Fear avoidance will be measured at baseline at 5 follow-ups (3,6,12,18 and 24 months)
  Fear avoidance will be assessed with Fear Avoidance Belief Questionnaire (FABQ).
Change from baseline Self-efficacy at 3,6,12,18 and 24 months assessed with Pain Self-Efficacy Questionnaire (PSEQ) | Self-efficacy will be measured at baseline at 5 follo-ups (3,6,12,18 and 24 months)
  Self-efficacy will be assessed with Pain Self-Efficacy Questionnaire (PSEQ)
Change from baseline Shoulder Function at 3,6,12,18 and 24 months assessed with Shoulder Pain and Disability Index (SPADI) | Function will be measured at baseline and 5 follow-ups (3,6,12,18 and 24 months)
  Function will be assessed with Shoulder Pain and Disability Index (SPADI)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Calderon J, Struyf F, Meeus M, Morales-Ascencio JM, Luque-Suarez A. Influence of psychological factors on the prognosis of chronic shoulder pain: protocol for a prospective cohort study. BMJ Open. 2017 Mar 6;7(3):e012822. doi: 10.1136/bmjopen-2016-012822. PMID 28264825